CLINICAL TRIAL: NCT02147860
Title: Full Day and Night Closed-Loop With DiAs Platform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Daniel Chernavvsky, MD, CRC, Prinicipal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17375; 2014PG-T1D038 (Other: The Leona M. & Harry B. Helmsley Charitable Trust Grant)
Record Dates: First submitted 2014-05-21; First posted 2014-05-28 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2015-11

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1; Artificial Pancreas Project (APP); Diabetes Assistant (DiAs); Closed-Loop Control (CLC); Continuous Glucose Monitor (CGM); Insulin Pump
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sensor Augmented Pump Therapy (Placebo Comparator): Each camp participant will be randomized to full day and night CLC or sensor augmented pump therapy for up to 7 days/6 nights. The subject will wear a continuous glucose monitoring system (CGM) to measure sensor glucose and a physiological monitor to measure heart rate and 3-axis accelerometer for 24-72 hours.
  Interventions: Other: Sensor Augmented Pump Therapy
- Diabetes Assistant (DiAs) with USS Virginia (Experimental): With the use of the UVA Artificial Pancreas (DiAs), the study will assess safety and feasibility and are not powered for statistical significance. These studies are intended to train staff on system function and obtain data regarding safe and feasible system use.
  Camp participants will be randomized to either closed-loop control using the DiAs or sensor-augmented pump therapy only. These studies would generate up to 120 days of closed-loop data and 120 comparable days of open-loop data.
  Interventions: Device: Diabetes Assistant (DiAs) with USS Virginia

INTERVENTIONS:
Device: Diabetes Assistant (DiAs) with USS Virginia — DiAs is the central component of our system. It is a standard cell phone running on an Android operating system. The cell phone has been changed to prevent from (1) using it as a phone or browser, (2) changing the volume (3) accidentally shutting it off. The cell phone runs an algorithm and is connected to work with the insulin pump and continuous glucose monitor to help keep the blood sugar in a desired range and help avoid hypoglycemia during the night.
  Other Names: Closed-Loop system
  Arms: Diabetes Assistant (DiAs) with USS Virginia
Other: Sensor Augmented Pump Therapy — Subjects randomized to this placebo group will wear a continuous glucose monitoring system (CGM) to measure sensor glucose and a physiological monitor to measure heart rate and 3-axis accelerometer for 24-72 hours.
  Other Names: SAP
  Arms: Sensor Augmented Pump Therapy

SUMMARY:
The overall aim of this proposed research is to determine the safety, feasibility and efficacy of the Diabetes Assistant (DiAs) controller in day and night closed-loop control in children and adolescents with type 1 diabetes over multiple days in a diabetes camp setting. This will be addressed in two parts: 1) An in residence, outpatient study to determine safety and feasibility of the DiAs during 72 continuous hours of day and night glucose control; and 2) Camp studies planned for the summer of 2014 with randomization to either full closed-loop or sensor-augmented pump therapy over the duration of 6-7 day diabetes camps.

DETAILED DESCRIPTION:
This study is an early feasibility study that will test the efficacy of DiAs - a smart-phone-based system compared to sensor augmented therapy in an outpatient setting. Twelve study subjects with type 1 diabetes, six each at UVa and Stanford University, who have experience with insulin pump use at two clinical sites will be recruited. The first six subjects recruited will be aged 15-18 years and this will follow with recruitment of six subjects aged 10-14 years. This study is designed to mimic the protocol at camp and will include a period of light exercise after breakfast and moderate intensity physical activity after lunch, with group activities such as soccer and volleyball. The duration of the Outpatient in Residence Study will be 72 hours. The data will be reviewed by the Data Safety Monitoring Board (DSMB) before proceeding to camp studies.

The camp study will recruit 48 subjects, with type 1 diabetes who have experience with insulin pump therapy. Initial studies will be conducted at a camp with older participants aged 15-35 years, with at least 5 of the campers between 15-18 years old. These studies will be reviewed by the DSMB and, if safe, we will recruit additional children aged 10-14 years of age. The duration of the Diabetes Camp Studies will be up to 7 days/6 nights.

ELIGIBILITY:
Inclusion Criteria: To be eligible for the study, a subject must meet the following criteria:

1. Clinical diagnosis of type 1 diabetes

   * The diagnosis of type 1 diabetes is based on the investigator's judgment
   * C peptide levels and antibody determinations are not required
2. Daily insulin therapy for ≥ 12 months
3. Insulin pump therapy for ≥ 3 months
4. Age 10.0 - 35.0 years
5. Avoidance of acetaminophen-containing medications (i.e. Tylenol) while wearing the continuous glucose monitor.
6. Willingness to wear a continuous glucose sensor and physiological monitor for the duration of the study
7. Female subjects who are sexually active must be on acceptable method of contraception (e.g. oral contraceptive pill, diaphragm, IUD)

Exclusion Criteria: The presence of any of the following is an exclusion for the study:

1. Diabetic ketoacidosis in the past month
2. Hypoglycemic seizure or loss of consciousness in the past 3 months
3. History of seizure disorder (except for hypoglycemic seizure)
4. History of any heart disease including coronary artery disease, heart failure, or arrhythmias
5. Cystic fibrosis
6. Current use of oral glucocorticoids, beta-blockers or other medications, which in the judgment of the investigator would be a contraindication to participation in the study.
7. History of ongoing renal disease (other than microalbuminuria).
8. Subjects requiring intermediate or long-acting insulin (such as NPH, Detemir or Glargine).
9. Subjects requiring other anti-diabetic medications other than insulin (oral or injectable).
10. Pregnancy - verbal denial of pregnancy obtained with telephone informed consent, pregnancy test performed at camp before study devices are assigned.
11. Sexually active females who do not practice acceptable contraceptive methods to prevent pregnancy.
12. Presence of a febrile illness within 24 hours of admission or acetaminophen use while wearing the CGM. The subject may be rescheduled for Research House/hotel admission if these criteria are not met. The camp study subject will not participate in the trial if these conditions are met.
13. Medical or psychiatric condition that in the judgment of the investigator might interfere with the completion of the protocol such as:

    * Inpatient psychiatric treatment in the past 6 months
    * Uncontrolled adrenal insufficiency
    * Alcohol abuse

Ages: 10 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2014-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
DiAs time within target | 7 days/6 nights
  Determine the efficacy of glucose control, as determined by the percentage of sensor glucose readings in the target range

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Buckingham, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - University of Virginia Center for Diabetes Technology, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Paper Published in Diabetes Care

REFERENCES:
- [Result] Ly TT, Buckingham BA, DeSalvo DJ, Shanmugham S, Satin-Smith M, DeBoer MD, Oliveri MC, Schertz E, Breton MD, Chernavvsky DR. Day-and-Night Closed-Loop Control Using the Unified Safety System in Adolescents With Type 1 Diabetes at Camp. Diabetes Care. 2016 Aug;39(8):e106-7. doi: 10.2337/dc16-0817. Epub 2016 Jun 6. No abstract available. PMID 27271182
- See also: Pubmed — http://www.ncbi.nlm.nih.gov/pubmed/?term=Chernavvsky+D